CLINICAL TRIAL: NCT05262842
Title: A Phase Ⅰ/Ⅰb Study to Investigate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of Toripalimab (Anti-PD-1 Antibody) in Combination With Senaparib (PARP Inhibitor) in Patients With Advanced Solid Tumors
Brief Title: JS001+IMP4297 in Patients With Advanced Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The sponsor voluntarily terminated the study before it was initiated
Sponsor: Shanghai Junshi Bioscience Co., Ltd. (Other)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS001-047-I
Record Dates: First submitted 2022-02-22; First posted 2022-03-02 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Intervention Model Description: Single Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS001+IMP4297 (Experimental)
  Interventions: Drug: JS001+IMP4297

INTERVENTIONS:
Drug: JS001+IMP4297 — Phase I: Dose Escalation The primary endpoints are the safety and tolerability of the combination, including the incidence and nature of DLTs and the determination of the MTD and RP2D. A 3 + 3 dose-escalation (60mg,80mg,100mg)design will be used. Patient in each dose level will be treated with toripalimab 240mg in combination with senaparib.
  Phase Ib: Dose Expansion This part will commence after the RP2D is determined and will further evaluate the safety and anti-tumor activity of toripalimab and senaparib in patients with specific types of advanced solid tumors. Patients will be enrolled concurrently into 5 exploratory cohorts with approximately 20 patients each cohort.

SUMMARY:
This is a Phase I/Ib open-label, multicenter study to evaluate the safety, tolerability, pharmacokinetics (PK), immunogenicity and antitumor activity of toripalimab in combination with senaparib in patients with advanced solid tumors. The study consists of 2 parts, the Phase I part of the study will be a dose-escalation evaluation to determine the RP2D of senaparib to be administered in combination with the fixed dose of toripalimab, and the Phase Ib portion will further evaluate the RP2D and evaluate the efficacy of combination in specific types of advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent and can understand and comply with the requirements of the study；
2. Male or female patients, age ≥ 18 years;
3. Patients with histologically or cytologically confirmed advanced (metastatic and/or unresectable) solid tumors that is incurable and have progressed during or after standard therapy or for which treatment is not available, or not tolerated;
4. Patients are able to provide fresh or archival tumor tissues (FFPE block or unstained slides). In the absence of archival tumor tissues, a fresh biopsy of a tumor lesion at baseline is recommended;
5. Patient must have at least one measurable lesion as defined per RECIST v1.1;
6. Eastern Cooperative Oncology Group (ECOG) Performalesce Status ≤1;
7. Life expectancy ≥12 weeks;
8. Vital organ function, defined as:

   Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L, hemoglobin ≥ 100 g/L.（Patients must not have required a blood transfusion or growth factor support ≤14 days before sample collection）； Serum creatinine ≤ 1.5 × upper limit of normal (ULN), or calculated creatinine clearance ≥ 51 mL/min using Cockcroft-Gault equation for patients with creatinine levels > 1.5×ULN； Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN, unless liver metastases are present, in which case they must be ≤ 5× ULN,ALP≤2.5 TIMES ULN (≤5 times ULN if tumor bone metastasis is present); Total bilirubin (TBIL) ≤ 1.5ULN; Patients with Gilbert syndrome should communicate with the sponsor medical examiner whether they can be enrolled in the group; Serum albumin ≥ 30 g/L； International standardized ratio (INR) or prothrombin time (PT) ≤ 1.5X ULN and activated partial thrombin time (aPTT) ≤ 1.5x ULN in patients who did not receive anticoagulant therapy; For those receiving anticoagulant therapy (e.g., low molecular weight heparin or warfarin), the anticoagulant dose should be stable for at least 4 weeks without dose adjustment; TSH within the normal range (if TSH is not within the normal range, free triiodothyronine (FT3) and free thyroxine (FT4) should be within the normal range.); Urinary protein -/+, if urinary protein ≥2+, additional 24-hour urine protein quantification test is required, such as 24-hour urine protein quantification <1g can be included in the group; Serum lipase or amylase ≤1.5 × ULN or >1.5 × ULN(no clinical or imaging confirmed pancreatitis); Fridericia's QT interval (QTc) prolongation: female≤ 470 ms, male≤ 450 ms at screening.
9. Ability to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening or otherwise altering the product formulation;
10. Toxicities of prior therapy (excepting alopecia) should be resolved to Grade≤ 1 as per Common Terminology Criteria for Adverse Event (CTCAE) v 5.0;
11. Females of reproductive age, and males whose partners are females of reproductive age, are required to use a medically approved contraceptive method (such as an intrauterine device (IUD), birth control pills or condoms) during and for 90 days after the study period; The serum HCG test of female patients of childbearing age must be negative within 7 days before study enrollment. And must be non lactation period;
12. For Phase Ib patients, the following requirements must be met:

Cohort A: Patients with recurrent or advanced endometrial cancer must meet the following criteria:

* Have progressed on or after platinum doublet therapy or intolerance to standard therapy
* Have received ≤ 2 prior lines of systemic therapies for recurrent or advanced disease. Patients may have received up to 1 additional line of chemotherapy if given in the neoadjuvant or adjuvant treatment setting, which may be concurrent or followed with chemoradiation).

Note: There is no restriction regarding prior hormonal therapy.

Cohort B: HRRm HER2-negative breast cancer patients with metastatic or locally advanced disease, which is unresectable, must meet the following criteria:

* For relapsed or advanced disease, progression follows systemic treatment of 0 to 3 lines; Hormone receptor positive (HR+) disease progressed on ≥1 endocrine therapy (adjuvant or metastatic), or not suitable, prior CDK 4/6i are allowed
* Patients must have documented evidence of a known deleterious or suspected deleterious germline orsomatic HRR gene mutations
* If patients have received platinum therapy, there should be:

In advanced setting: no evidence of objective disease progression while receiving platinum In (neo-)adjuvant setting: disease-free interval of ≥6 months after the last dose

Cohort C: Patients with small cell lung cancer (SCLC) must meet the following criteria:

• Extensive small-cell lung cancer (according to the American Veterans Lung Cancer Association VALG stage) with progression on or intolerance to standard therapy

Cohort D: Patients with recurrent or advanced stage III B-C or IV (AJCC Version 8) NSCLC must meet the following criteria:

* No known EGFR-sensitising mutations and ALK fusion, testing is not mandatory for patients with squamous cell cancer
* 1)PD-L1 TPS≥1%, has not received any prior systemic antitumor therapy.Prior use of neoadjuvant and/or adjuvant antitumor therapy is permitted provided that the time between the end of the (new) adjuvant therapy and the onset of recurrence/metastasis is ≥6 months. Or 2) Have progressed after at least 1 prior systemic therapy for recurrent or advanced disease or intolerance to standard thera, first-line use of PD-1/PD-L1 inhibitors (either monotherapy or combination chemotherapy) is allowed, but those who have previously received PARP inhibitors cannot be included.

Cohort E: Other tumor types that may carry DNA damage repair defects that are sensitive to PARP inhibitors or ikely to be responsive to PD-L1/PD-1 inhibitors,including but not limited to, advanced or metastatic nasopharyngeal carcinoma, recurrent epithelial ovarian cancer, metastatic castration-resistant prostate cancer, locally advanced or metastatic urothelial carcinoma (muscular-invasive bladder cancer, ureteral cancer, urethral or pelvic cancer), and advanced or metastatic pancreatic adenocarcinoma.

Exclusion Criteria:

1. Major surgery (as defined by the investigator) within 4 weeks of starting study treatment and patient must have recovered from any effects of any major surgery; Note: Local palliative treatment (eg. local surgery or radiotherapy) for isolated lesions is allowed, if not affecting the efficacy evaluation;
2. Patient has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Patients with spinal cord compression unless considered to have received definitive treatment for this and evidence of clinically stable disease for 4 weeks; Note: Patients with previously treated brain metastases may participate provided they are stable and have no symptoms.Asymptomatic patients with brain metastases found at screening phase are eligible.Carcinomatous meningitis precludes a patient from study participation regardless of clinical stability.
3. Patient has an active autoimmune disease or autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

   Note: ① Autoimmune diseases include but are not limited to systemic lupus erythematosus, interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism or multiple sclerosis; ② patients with vitiligo or in childhood asthma has complete remission, adult patients without any intervention can be incorporated into; ③ in chronic obstructive pulmonary disease (COPD), asthma need continuous use of bronchiectasis, inhaled corticosteroids, or local injection of corticosteroids can into the group of patients.
4. Prior malignancy within the previous 5 years except for locally curable cancers that have apparently been cured (eg, basal or squamous cell skin cancer, or carcinoma in situ of the cervix, breast);
5. Patient is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease. Specific examples include, but are not limited to, uncontrolled hypertension (systolic blood pressure >160 mmHg, diastolic blood pressure >100 mmHg); recent (within 90 days) NYHA≥3 heart failure, unstable angina, unstable arrhythmia, myocardial infarction or cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism; LVEF<50%;; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent);
6. Severe chronic or active infections (including tuberculosis infection, etc) requiring systemic antibacterial, antifungal, or antiviral therapy within 14 days prior to first dose of study drugs; Patients with active tuberculosis (TB) who are receiving anti-TB treatment or have received anti-TB treatment within 1 year prior to screening;
7. Patients who have a history of or are currently developingpneumonitisrequiring steroid treatment, including but not limited to interstitial pneumonia, radiation pneumonia, pulmonary fibrosis, or machine-induced pneumonia;
8. Prior bone marrow allogeneic transplantation or solid organ transplantation;
9. Patient has any known history of MDS/AML or a pre-treatment cytogenetic testing result at risk for a diagnosis of MDS/AML;
10. Patients who had prior therapy of an anti-PD-1, anti-PD-L1, anti-PD-L2（SCLC and NSCLC cohorts were excluded） or prior treatment with a PARPi；
11. Patient is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy within 4 weeks of the first dose of treatment;
12. Prior chemotherapy or other systemic anticancer therapy (eg, targeted therapy) within 4 weeks prior to start of study treatment; 6 weeks for nitrosoureas or mitomycin. Hormonal therapy for cancer treatment is allowed until 7 days prior to study treatment. Any herbal medicine used to control cancer within 14 days of the first study treatment;
13. Requirement for systemic treatment with corticosteroids or other immunosuppressive medications within 2 weeks of study drug administration. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection), or systemic corticosteroids at physiologic doses (prednisone≤10 mg/day or its equivalent), or steroids as premedication for hypersensitivity reactions (eg, contrast agent allergy) are allowed;
14. Concomitant use of known strong cytochrome CYP3A4 inhibitors (eg, itraconazole, telithromycin, clarithromycin, protease inhibitors boosted with ritonavir or cobicistat, indinavir, saquinavir, nelfinavir, boceprevir, telaprevir). The required washout period prior to starting senaparib is 2 weeks;
15. Concomitant use of known strong CYP3A4 inducers (eg, phenobarbital, enzalutamide, phenytoin, rifampicin, rifabutin, rifapentine, carbamazepine, nevirapine and St John's Wort) . The required washout period prior to starting senaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents;
16. Use of live attenuated vaccines within 30 days of initiation of study therapy; Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP；
17. Patients known to have active hepatitis (i.e., hepatitis B or C) or humales immunodeficiency virus (HIV) positive:

    * Hepatitis B core antibody (HBcAb) positive and hepatitis B surface antigen (HBsAg) negative during screening period can participate in this study; Before enrollment, such patients must be tested for HBV DNA, whose HBV DNA is less than the lower limit of detection before enrollment;
    * Subjects who are HBsAg positive and whose HBV DNA is below the test threshold can be enrolled, assessed by the investigator at risk, and treated with anti-HBV therapy to avoid viral activation throughout the study, if necessary;
    * Patients with positive hepatitis C virus (HCV) antibodies can only be enrolled if the HCV RNA test results are negative
18. Patient has a known hypersensitivity to senaparib or toripalimab components or excipients;
19. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-03-29 (Estimated); Primary Completion 2024-04-06 (Estimated); Study Completion 2024-06-06 (Estimated)

PRIMARY OUTCOMES:
DLT、AE、SAE、irAE | 3 years
  Safety endpoints: incidence and severity of DLT, adverse events (AE), serious adverse events (SAE), and immune-related adverse events (irAE); Abnormal changes in laboratory and other tests with clinical significance
MTD | 1 year
  Maximum tolerated dose (MTD)
RP2D | 1 year
  Recommended dose for phase II trial
ORR | 2 years
  Efficacy endpoints: Objective response rate (ORR) per RECIST v1.1

SECONDARY OUTCOMES:
DOR | 2 years
  Efficacy endpoints: Duration of response (DOR) per RECIST v1.1
DCR | 2 years
  Efficacy endpoints: Disease control rate (DCR) per RECIST v1.1
PFS | 2 years
  Efficacy endpoints: Progression-free survival (PFS) per RECIST v1.1
OS | 2 years
  Efficacy endpoints: Overall survival (OS)
Pharmacokinetic (PK) characteristics | 2 years
  Drug concentration of individual subjects at different time points after administration
Peak concentration（Cmax） | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：peak concentration (Cmax) ;
Peak time（Tmax） | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：peak time (Tmax) ;
Valley concentration（Ctrough） | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：valley concentration（Ctrough）；
Area under blood concentration-time curve (AUC0-tand AUC0-inf) | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：area under blood concentration-time curve (AUC0-tand AUC0-inf) ;
Volume of distribution (Vss) | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：volume of distribution (Vss)
Elimination half-life (T1/2) and other parameters | 2 years
  The pharmacokinetic parameters of JS002 and Toripalimab (JS001) ：elimination half-life (T1/2) and other parameters
Clearance rate (CL) | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：clearance rate (CL) ;
Mean retention time（MRT） | 2 years
  The pharmacokinetic parameters of IMP4297 and Toripalimab (JS001) ：mean retention time（MRT）
ADA against | 2 years
  The incidence of ADA and/or neutralizing antibody (Nab), ADA titer;

OTHER OUTCOMES:
Correlation between biomarkers and clinical efficacy | 2 years
  Biomarker assessments, including but not limited to PD-L1 expression, TMB, and gene expression profiling

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, M.D., Principal Investigator — Sun Yat-sen University

IPD SHARING:
Plan to Share IPD: No